CLINICAL TRIAL: NCT04238286
Title: Analgesic Efficacy of Dry Needling in Fibromyalgia Patients.Influence of Catastrophism in the Successful Intervention
Brief Title: Influence of Catastrophism in Fibromyalgia Patients Following Dry Needling Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Collaborators: Fundación Universidad Católica de Valencia San Vicente Mártir (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: U1111-1242-5849 (UTN)
Record Dates: First submitted 2020-01-20; First posted 2020-01-23 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Myofascial Pain Syndrome; Catastrophizing; Chronic Pain
Keywords: Fibromyalgia; Female; Myofascial trigger points
MeSH Terms: conditions — Myofascial Pain Syndromes; Chronic Pain; Fibromyalgia | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dry needling group (Experimental): Patients treated with dry needling
  Interventions: Procedure: Dry needling
- Sham group (Sham Comparator): Patients treated with a simulated dry needling
  Interventions: Procedure: Dry needling
- Control (No Intervention): Patients never treated

INTERVENTIONS:
Procedure: Dry needling — All the participants will be placed in a prone position on the bench. Once the subject is settled, we will localize a nodule within the palpable taut band, confirming its presence after inducing local twitch response by palpation. After placing the MTrPs, the area will be sterilized with an alcohol solution colorless spray [Skin-des. Agupunt ®]. The puncture method used in the true dry needling groups will be the Hong's fast in-fast out technique, described as the most aggressive technique in the MTrPs treatment, using a needle of 0.32 x 40 mm. The intervention will be implemented until the subject reports the presence of seven local twitch reactions to the controller.
  Arms: Dry needling group; Sham group

SUMMARY:
Background: Dry needling trigger point treatment, while painful, has been demonstrated as a useful tool in fibromyalgia patients for decreasing pain and central sensitization. However, the current biopsychosocial pain paradigm indicates that fibromyalgia subjects with high levels of catastrophizing have negative thoughts related with perceived partner responses to pain, which results in an emotional and physical stress after a painful episode.

Objective: To assess whether catastrophizing could influence the perception of pain during and after dry needling application.

Study design: A singled-blind randomized controlled trial.

Setting: Department of Medicine, Faculty of Health Sciences, Universitat Jaume I

Methods: Female fibromyalgia patients and number and age-matched female controls will be recruited and randomly assigned to either a real or a simulated dry needling group. The Spanish version of the pain catastrophizing scale will be used to assess the catastrophizing level of each participant before initiating any of the planned interventions. The perceived pain during and immediately after the dry needling procedure will be measured using the pain visual analogue scale, [VAS].

DETAILED DESCRIPTION:
Fibromyalgia syndrome (FS) is currently classified as chronic widespread pain with widespread allodynia (Coster et al., 2008). These symptoms are accompanied by other disorders, such as sleep disturbance, headaches, morning stiffness, irritable bowel syndrome, interstitial cystitis, dyspareunia, mood disturbances and depression (Gerwin, 2005). The World Health Organization recognized FS as a disease in 1992, basing its decision on the diagnostic criteria of the American College of Rheumatology (ACR) which has recently been criticized and updated (Wolfe et al., 2011; Wolfe et al., 2010; Wolfe and Hauser, 2011). Depending on the diagnostic criteria used, the prevalence is from 2% to 8% of the population increasing with age, with highest values attained between 60 and 70 (Stahl, 2009). In Spain, was estimated that 2.4% of the population over 20 years old presents the disease, and it is higher in females than in males (ratio 21:1) (Cordero, 2011).

A central sensitivity syndrome could be the most plausible explanation for chronic widespread pain affecting people with fibromyalgia syndrome. Although it was suggested this condition was the sole cause (Yunus, 2007), central sensitization of the nervous system causes the phenomena of hyperalgesia and allodynia in the individual suffering from chronic pain (Butler and Moseley, 2003) .

The subject with chronic pain has an altered alarm system; this alteration could be initiated by a peripheral sensitization (Sarzi-Puttini et al., 2011) activated by the release of various chemical substances such as substance P, serotonin and bradykinin (Yunus, 2007). Myofascial trigger points (MTrPs) are able to maintain this peripheral sensitization (Affaitati et al., 2011; Ge et al., 2010) by triggering the spontaneous pain patterns experienced by a patient with fibromyalgia syndrome (Ge et al., 2011).

MTrPs contain algogenic substances capable of generating changes in the intensity of pain. Differences in the concentration of these substances between healthy muscle and MTrPs (Shah et al., 2005) have been shown. One of the most effective techniques for the treatment of MTrPs is dry needling (Mayoral, 2010), because it alters the chemical environment of the MTrPs, thus decreasing their sensitization (Dommerholt, 2011). However, there are as until no few studies that have examined the effectiveness of this technique in patients with FS (Chou et al., 2008; Staud, 2006). Moreover, in these patients the perception of pain during and after treatment can be influenced not only by central sensitization, but also by psychosocial variables.

Catastrophization, considered to be the basic psychological construction concerning the perception of pain intensity, is a cognitive and emotional process encompassing magnification of pain-related stimuli, feelings of helplessness, and a generally pessimistic orientation (Labus et al., 2003; Rodero et al., 2010). This catastrophization, understood as a set of negative emotions and cognitive processes, is a risk factor in fibromyalgia and leads to an increase in symptoms, health status warning, symptoms of helplessness and pessimism (Alegre de Miquel and Sellas Fernandez, 2008; Sullivan et al., 2001).

These negative thoughts lead to alterations in the function of the descending inhibitory pathways that modulate pain (Wideman and Sullivan, 2011) producing an increase in the pain's intensity and exaggerated pain behavior (Wideman and Sullivan, 2012). Several lines of research suggest that this psychological construct is an indicator of poor results obtained from various treatments (surgical, pharmacological and psychological interventions in pain management) (Sullivan et al., 2009; Mankovsky et al., 2012; Sullivan et al., 2005).

Catastrophizing is an important factor in the pathophysiological FM, which also influences the perception of pain and the effects of the various treatments mentioned above. Several studies have shown that catastrophizing increases attention at the site of injury and increases the fear of pain that patient refers (McMahon et al., 2013; Sullivan et al., 2001). However, how this psychological construct may influence both factors - the treatment effectiveness of MTrPs by dry needling and the perception of pain during this treatment - is still unknown.

Subjects who experience high levels of catastrophizing have been demonstrated as having increased emotional and physical stress in response to a painful episode. It would therefore be interesting to analyze whether high levels of catastrophizing may influence and be related with high levels of perceived pain during and after dry needling treatment.

The main objective of our study is to assess whether catastrophizing could influence the perception of pain during and after dry needling application.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of fibromyalgia verified by a qualified rheumatologist according to the ACR criteria
* To have basic spanish skills (be able to understand oral and written spanish language)

Exclusion Criteria:

* Belonephobia or mimicking pathologies
* Lymphedema
* Pregnancy
* Neoplastic disorders

Ages: 35 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Although the condition affects both sexes, women are far more likely to develop fibromyalgia.
Enrollment: 120 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
The Pain Catastrophizing Scale (PCS) is a 13-item self-administered scale and one of the most widely used to assess pain catastrophizing | 48 hours
  The theoretical range of the instrument is between 0 and 52, with low scores indicating low catastrophizing, and high values showing high catastrophizing. Compare to others this questionnaire is unique since the individual does not need to be in pain while completing it.

SECONDARY OUTCOMES:
Pain Intensity Measure VAS | 48 hours
  The pain visual analogue scale [VAS] is designed to provide a broad and comprehensive assessment, albeit a subjective one, of the pain dimensions. A visual analogue scale is a straight vertical or horizontal line, the length of which represents the continuum of the painful experience. It consists of a 10 cm horizontal line, with perpendicular lines at the ends representing the inner and outer limits of the measured pain construct. The anchor points at each end point are characterized by a brief verbal expression such as 'nothing' or 'no pain' at one end and "unbearable" at the other. Verbal descriptors are usually accompanied by a number [e.g., "nothing" can be accompanied by 0 and "unbearable" by 10].
Algometry | 48 hours
  Measurement of pain by means of an algometer, an instrument for determining sensitivity to pain produced by pressure (Kg/cm2).

CONTACTS AND LOCATIONS:
Overall Officials: Juan Vicente Mampel, PhD, Principal Investigator — Universidad Catolica San Vicente Martir
Locations (1):
- Universitat Jaume I, Castellon, Castellón, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ge HY, Fernandez-de-Las-Penas C, Madeleine P, Arendt-Nielsen L. Topographical mapping and mechanical pain sensitivity of myofascial trigger points in the infraspinatus muscle. Eur J Pain. 2008 Oct;12(7):859-65. doi: 10.1016/j.ejpain.2007.12.005. Epub 2008 Jan 18. PMID 18203637
- [Result] Sullivan M, Tanzer M, Stanish W, Fallaha M, Keefe FJ, Simmonds M, Dunbar M. Psychological determinants of problematic outcomes following Total Knee Arthroplasty. Pain. 2009 May;143(1-2):123-9. doi: 10.1016/j.pain.2009.02.011. Epub 2009 Mar 21. PMID 19304392
- [Result] Sarzi-Puttini P, Atzeni F, Mease PJ. Chronic widespread pain: from peripheral to central evolution. Best Pract Res Clin Rheumatol. 2011 Apr;25(2):133-9. doi: 10.1016/j.berh.2011.04.001. PMID 22094190
- [Result] Affaitati G, Costantini R, Fabrizio A, Lapenna D, Tafuri E, Giamberardino MA. Effects of treatment of peripheral pain generators in fibromyalgia patients. Eur J Pain. 2011 Jan;15(1):61-9. doi: 10.1016/j.ejpain.2010.09.002. PMID 20889359